CLINICAL TRIAL: NCT06744673
Title: A Retrospective, Observational Study Using a Healthcare Database to Assess the Pregnancy Outcome in Women Exposed to Dayvigo® During Pregnancy Compared to an Unexposed Control Population
Brief Title: A Study to Assess the Pregnancy Outcome in Women Exposed to Dayvigo® During Pregnancy Compared to an Unexposed Control Population
Status: Active, not recruiting | Type: Observational
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: E2006-A001-604
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Sleep Initiation and Maintenance Disorders; Pregnancy
Keywords: Insomnia; Pregnancy; Dayvigo; Lemborexant; E2006
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort A: Dayvigo-exposed Cohort: Pregnant women participants with a diagnosis of insomnia within the 6 months before the estimated date of conception (DOC) and who have received at least 1 dose of Dayvigo at any time from 10 days after the last menstrual period (LMP) that is, 4 days prior to the DOC, which is 5 times the product's half-life, until the pregnancy outcome (that is, any trimester) will be observed retrospectively.
  Interventions: Other: No Intervention
- Cohort B: Comparator-exposed Cohort: Pregnant women participants with a diagnosis of insomnia within the 6 months before the estimated DOC and who have received at least 1 dose of drug indicated for the treatment of insomnia other than Dayvigo from 5 times the product's half-life prior to the estimated DOC until the pregnancy outcome, and no exposure to Dayvigo between 10 days after the LMP and the pregnancy outcome (that is, any trimester) will be observed retrospectively.
  Interventions: Other: No Intervention
- Cohort C: Untreated Unexposed Comparator Cohort: Pregnant women participants with a diagnosis of insomnia within the 6 months before the estimated DOC and who were not exposed to any prescribed medication for the treatment of insomnia during pregnancy, that is, from 5 times the product's half-life prior to the estimated DOC until the pregnancy outcome (that is, any trimester) will be observed retrospectively.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
The primary purpose of the study is to compare the occurrence of major congenital malformations (MCMs) among live births between women with insomnia who are exposed to Dayvigo during the 1st trimester of pregnancy and women with insomnia who are not exposed to any prescription insomnia drugs at any time during the pregnancy and to compare the occurrence of MCMs among live births between women with insomnia who are exposed to Dayvigo during the 1st trimester of pregnancy and women with insomnia who are exposed to a prescription insomnia drug other than Dayvigo during the 1st trimester of pregnancy.

DETAILED DESCRIPTION:
As this is a Retrospective Database study, the Study Start Date for this study references the date at which data will become available

ELIGIBILITY:
Inclusion Criteria:

1. Must be female.
2. Must be 16 to 49 years of age
3. Has a clinically recognized pregnancy that overlaps with the data collection period between 01 Jun 2020 and the end of the data collection period
4. Has continuous medical and pharmacy benefit coverage for a minimum of 6 months (Baseline Period) before the estimated date of conception and through the date of pregnancy outcome.

Cohort A:

1. Exposed to at least 1 dose of Dayvigo at any time from 10 days after the LMP, that is, approximately 4 days prior to the estimated DOC, defined as 14 days after the LMP, based on the product's half-life, until the pregnancy outcome
2. Has a diagnosis of insomnia recorded in her electronic healthcare data within 6 months before the estimated DOC, insomnia defined as an International Classification of Disease (ICD) 10-CM code G47.0x Insomnia or ICD 10 CM code F51.0x Insomnia not due to a substance or known physiological condition or Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) code 780.52. Or if the first exposure to Dayvigo occurs after the DOC, then must have a diagnostic code for insomnia prior to or on the first exposure to this drug.

Cohort B:

1. Exposed to at least 1 dose of prescription medication for insomnia other than Dayvigo from 5 times the product's half-life prior to the estimated DOC until the pregnancy outcome (that is, any trimester)
2. Has a diagnosis of insomnia recorded in her electronic healthcare data within 6 months before the estimated DOC, insomnia defined as an ICD 10-CM code G47.0x Insomnia or ICD 10 CM code F51.0x Insomnia not due to a substance or known physiological condition or DSM-5 code 780.52. Or if the first exposure to the prescription insomnia medication occurs after the DOC, then must have a diagnostic code for insomnia prior to or on the first exposure to this drug

Cohort C:

1. Not exposed to any prescription medication for the treatment of insomnia during pregnancy that is, from 5 times the product's half-life prior to the estimated DOC until the pregnancy outcome (that is, any trimester). NB: May be exposed during pregnancy to other drugs (that is, not for insomnia), but only provided that these are not associated with potential or known teratogenicity
2. Has a diagnosis of insomnia recorded in her electronic healthcare data within 6 months before the estimated DOC, insomnia defined as an ICD 10-CM code G47.0x Insomnia or ICD 10 CM code F51.0x Insomnia not due to a substance or known physiological condition or DSM-5 code 780.52

Exclusion Criteria:

1. Identified pregnancies with exposure to known teratogens during pregnancy, that is, from 14 days after the LMP to pregnancy outcome (any trimester) or to dual orexin receptor antagonists other than lemborexant (this includes, but it is not limited to, exclusion of suvorexant and daridorexant) from 5 times the product's half-life prior to the estimated DOC until the pregnancy outcome (any trimester) will be excluded
2. Pregnancies not associated with a known pregnancy outcome.

Ages: 16 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: The study population will include pregnant women with insomnia.
Sampling Method: Non-Probability Sample
Enrollment: 861 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Live Births Reported With MCM in Women of Cohort A Subset and Cohort C | At estimated date of delivery (EDD)/pregnancy outcome (up to 1 year 10 months)
  MCM will be defined as an abnormality of body structure or function that is present at birth, is of prenatal origin (that is, birth defect), has significant medical, social, or cosmetic consequences for the affected individual, and typically requires medical intervention. Congenital anomalies will be classified using the Centers for Disease Control and Prevention (CDC)'s Metropolitan Atlanta Congenital Defects Program (MACDP) system. Live birth will be defined as birth of a living fetus at greater than or equal to (>=) 20 gestational weeks or, if gestational age is unknown, a fetus weighing >=350 grams (g). Cohort A subset is defined as women with insomnia who are exposed to Dayvigo during the 1st trimester of pregnancy.
Percentage of Live Births Reported With MCM in Women of Cohort A and Cohort B Subsets | At EDD/pregnancy outcome (up to 1 year 10 months)
  MCM will be defined as an abnormality of body structure or function that is present at birth, is of prenatal origin (that is, birth defect), has significant medical, social, or cosmetic consequences for the affected individual, and typically requires medical intervention. Cohort A subset is defined as women with insomnia who are exposed to Dayvigo during the 1st trimester of pregnancy and Cohort B subset is defined as women with insomnia who are exposed to a prescription insomnia drug other than Dayvigo during the 1st trimester of pregnancy.

SECONDARY OUTCOMES:
Percentage of Live Births and Fetal Losses With MCM in Women of Cohort A and Cohort B Subsets | At EDD/pregnancy outcome (up to 1 year 10 months)
  MCM will be defined as an abnormality of body structure or function that is present at birth, is of prenatal origin (that is, birth defect), has significant medical, social, or cosmetic consequences for the affected individual, and typically requires medical intervention. Congenital anomalies will be classified using the CDC's MACDP system. Live birth will be defined as birth of a living fetus at >=20 gestational weeks or, if gestational age is unknown, a fetus weighing >=350 g. Cohort A subset is defined as women with insomnia who are exposed to Dayvigo during the 1st trimester of pregnancy and Cohort B subset is defined as women with insomnia who are exposed to a prescription insomnia drug other than Dayvigo during the 1st trimester of pregnancy.
Percentage of Live Births and Fetal Losses With MCM in Women of Cohort A Subset and Cohort C | At EDD/pregnancy outcome (up to 1 year 10 months)
  MCM will be defined as an abnormality of body structure or function that is present at birth, is of prenatal origin (that is, birth defect), has significant medical, social, or cosmetic consequences for the affected individual, and typically requires medical intervention. Congenital anomalies will be classified using the CDC's MACDP system. Live birth will be defined as birth of a living fetus at >=20 gestational weeks or, if gestational age is unknown, a fetus weighing >=350 g. Cohort A subset is defined as women with insomnia who are exposed to Dayvigo during the 1st trimester of pregnancy.
Percentage of Participants With Spontaneous Abortion (SAB) in Cohort A and Cohort B Subsets | From enrollment up to pregnancy outcome (up to 1 year 10 months)
  SAB is defined as an involuntary fetal loss or the expulsion of the products of conception occurring at less than (<) 20 gestational weeks. Cohort A subset is defined as women with insomnia who are exposed to Dayvigo during the 1st trimester of pregnancy and Cohort B subset is defined as women with insomnia who are exposed to a prescription insomnia drug other than Dayvigo during the 1st trimester of pregnancy.
Percentage of Participants With SAB in Cohort A Subset and Cohort C | From enrollment up to pregnancy outcome (up to 1 year 10 months)
  SAB is defined as an involuntary fetal loss or the expulsion of the products of conception occurring at <20 gestational weeks. Cohort A subset is defined as women with insomnia who are exposed to Dayvigo during the 1st trimester of pregnancy.
Percentage of Participants With Stillbirth in Cohort A and Cohort B Subsets | From 20 gestational weeks up to pregnancy outcome (up to 1 year 10 months)
  Stillbirth is defined by the American College of Obstetricians and Gynecologists (ACOG), an involuntary fetal loss occurring at >=20 gestational weeks or, if gestational age is unknown, a fetus weighing >=350 g. Cohort A subset is defined as women with insomnia who are exposed to Dayvigo during the 1st trimester of pregnancy and Cohort B subset is defined as women with insomnia who are exposed to a prescription insomnia drug other than Dayvigo during the 1st trimester of pregnancy.
Percentage of Participants With Stillbirth in Cohort A Subset and Cohort C | From 20 gestational weeks up to EDD/ pregnancy outcome (up to 1 year 10 months)
  Stillbirth is defined by the ACOG, an involuntary fetal loss occurring at >=20 gestational weeks or, if gestational age is unknown, a fetus weighing >=350 g. Cohort A subset is defined as women with insomnia who are exposed to Dayvigo during the 1st trimester of pregnancy.
Percentage of Participants With Preterm Birth in Cohort A and Cohort B Subsets | From enrollment up to pregnancy outcome (up to 1 year 10 months)
  Preterm birth is defined as a live birth occurring at <37 gestational weeks. Cohort A subset is defined as women with insomnia who are exposed to Dayvigo during the 1st trimester of pregnancy and Cohort B subset is defined as women with insomnia who are exposed to a prescription insomnia drug other than Dayvigo during the 1st trimester of pregnancy.
Percentage of Participants With Preterm Birth in Cohort A Subset and Cohort C | From enrollment up to pregnancy outcome (up to 1 year 10 months)
  Preterm birth is defined as a live birth occurring at <37 gestational weeks. Cohort A subset is defined as women with insomnia who are exposed to Dayvigo during the 1st trimester of pregnancy.
Percentage of Participants With Induced Termination in Cohort A and Cohort B Subsets | From enrollment up to date of induced termination (up to 1 year 10 months)
  Induced termination is defined as a pregnancy terminated according to the participant's decision (elective termination), with or without medical or therapeutic indication (therapeutic indication occurs when the pregnancy endangers the mother's health or the fetus has a condition incompatible with normal life). Cohort A subset is defined as women with insomnia who are exposed to Dayvigo during the 1st trimester of pregnancy and Cohort B subset is defined as women with insomnia who are exposed to a prescription insomnia drug other than Dayvigo during the 1st trimester of pregnancy.
Percentage of Participants With Induced Termination in Cohort A Subset and Cohort C | From enrollment up to date of induced termination (up to 1 year 10 months)
  Induced termination is defined as a pregnancy terminated according to the participant's decision (elective termination), with or without medical or therapeutic indication (therapeutic indication occurs when the pregnancy endangers the mother's health or the fetus has a condition incompatible with normal life). Cohort A subset is defined as women with insomnia who are exposed to Dayvigo during the 1st trimester of pregnancy.
Percentage of Infants With Small for Gestational Age (SGA) in Cohort A and Cohort B Subsets | At EDD/pregnancy outcome (up to 1 year 10 months)
  SGA will be evaluated as weight at birth in <10th percentile for sex and gestational age using standard growth charts for full and preterm live-born infants. Cohort A subset is defined as women with insomnia who are exposed to Dayvigo during the 1st trimester of pregnancy and Cohort B subset is defined as women with insomnia who are exposed to a prescription insomnia drug other than Dayvigo during the 1st trimester of pregnancy.
Percentage of Infants With SGA in Cohort A Subset and Cohort C | At EDD/pregnancy outcome (up to 1 year 10 months)
  SGA will be evaluated as weight at birth in <10th percentile for sex and gestational age using standard growth charts for full and preterm live-born infants. Cohort A subset is defined as women with insomnia who are exposed to Dayvigo during the 1st trimester of pregnancy.
Percentage of Live Births and Fetal Losses With MCM in Women of Cohort A, B and C | At EDD/pregnancy outcome (up to 1 year 10 months)
  MCM will be defined as an abnormality of body structure or function that is present at birth, is of prenatal origin (that is, birth defect), has significant medical, social, or cosmetic consequences for the affected individual, and typically requires medical intervention. Congenital anomalies will be classified using the CDC's MACDP system. Live birth will be defined as birth of a living fetus at >=20 gestational weeks or, if gestational age is unknown, a fetus weighing >=350 g.
Percentage of Participants With SAB in Cohort A, B and C | From enrollment up to pregnancy outcome (up to 1 year 10 months)
  SAB is defined as an involuntary fetal loss or the expulsion of the products of conception occurring at less than (<) 20 gestational weeks.
Percentage of Participants With Stillbirth in Cohort A, B and C | From 20 gestational weeks up to EDD/ pregnancy outcome (up to 1 year 10 months)
  Stillbirth is defined by the ACOG, an involuntary fetal loss occurring at >=20 gestational weeks or, if gestational age is unknown, a fetus weighing >=350 g.
Percentage of Participants With Preterm Birth in Cohort A, B and C | From enrollment up to pregnancy outcome (up to 1 year 10 months)
  Preterm birth is defined as a live birth occurring at <37 gestational weeks.
Percentage of Participants With Induced Termination in Cohort A, B and C | From enrollment up to date of induced termination (up to 1 year 10 months)
  Induced termination is defined as a pregnancy terminated according to the participant's decision (elective termination), with or without medical or therapeutic indication (therapeutic indication occurs when the pregnancy endangers the mother's health or the fetus has a condition incompatible with normal life).
Percentage of Infants With SGA in Cohort A, B and C | At EDD/pregnancy outcome (up to 1 year 10 months)
  SGA will be evaluated as weight at birth in <10th percentile for sex and gestational age using standard growth charts for full and preterm live-born infants.
Number of MCM From Postmortem With Non-live Birth in Cohort A and Cohort B | From enrollment up to pregnancy outcome (up to 1 year 10 months)
  Any findings of MCMs from postmortem examination of pregnancies with non-live birth outcomes (that is, abortions, fetal deaths/stillbirths) will be reported separately.

CONTACTS AND LOCATIONS:
Locations (1):
- Eisai Trial Site #1, Nutley, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.